CLINICAL TRIAL: NCT04219046
Title: Evaluation of Naloxegol, a Peripherally Acting µ-opioid Receptor Antagonist, in the Prevention of Postoperative Ileus After Cystectomy
Brief Title: Evaluation of Naloxegol in the Prevention of POI After Cystectomy
Acronym: ANTAGOCYST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANTAGOCYST-01-IPC 2019-034
Record Dates: First submitted 2019-12-20; First posted 2020-01-06 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer; Cystostomy; Complications
Keywords: Radical cystectomy; Postoperative ileus; Enhanced Recovery After Surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — naloxegol

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): ERAS program with administration of experimental treatment: Naloxegol 25mg administrated once daily from surgery for up to 7 days
  Interventions: Drug: Naloxégol oxalate
- Placebo (Placebo Comparator): ERAS program with administration of placebo: Placebo administrated once daily from surgery for up to 7 days
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Naloxégol oxalate — Oral administration once daily
  Other Names: Naloxegol
  Arms: Experimental Treatment
Drug: Placebo oral tablet — Oral administration once daily
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Postoperative ileus (POI) is defined as a transient reduction of bowel motility that prevents effective transit of bowel content and tolerance of oral intake following surgical interventions, especially after radical cystectomy. It remains a major factor associated with postoperative morbidity, length of hospital stay and medical costs.

In order to optimize perioperative care for patients undergoing radical cystectomy in a context of an ERAS (Enhanced Recovery After Surgery) program, we will evaluate the effectiveness of systemic pharmacologic opioid antagonist treatment.

DETAILED DESCRIPTION:
Radical cystectomy (RC) with urinary diversion represents the gold standard treatment for muscle-invasive bladder cancer. Postoperative ileus (POI) is defined as a transient reduction of bowel motility that prevents effective transit of bowel content and tolerance of oral intake following surgical interventions, especially after RC. It remains a major factor associated with postoperative morbidity, length of hospital stay and medical costs.

Faster gastrointestinal recovery and prevention of POI are at the heart of ERAS (Enhanced Recovery After Surgery) protocols. In order to optimize the post-operative consequences of patients operated on for a cystectomy within the framework of a RAAC program, several provisions aim to alleviate post-operative gastrointestinal dysfunctions.

Naloxegol, peripherally acting µ-opioid receptor antagonist, is currently approved for opioid-induced constipation in Chronic Non-Cancer Pain, but its potential interest to prevent POI has never been assessed. In this randomized, double-blind, placebo-controlled trial, the administration of Naloxegol for a limited duration as part of ERAS (Enhanced Recovery After Surgery) program will be evaluated to reduce the time of hospital discharge (length of stay) and to reduce the rate of postoperative complications. Priamry and secondary objectives will be compared between naloxegol and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Informed consent signed
* Histopathological confirmation of bladder cancer
* Patients undergoing radical cystectomy and urinary diversion for an oncological indication
* Patients able to understand the study procedures, agreed to participate in the study program
* Patients affiliated to the national "Social Security" regimen or beneficiary of this regimen

Exclusion Criteria:

* Unwilling to undergo cystectomy
* Cystectomy for non-oncological indication
* Patients with concomitant upper urinary tract disease
* Previous total colectomy, gastrectomy, or gastric bypass, or functional colostomy or ileostomy
* Previous pelvic radiotherapy for prostate or bladder cancer
* Patients having taken opioids for more than seven days before surgery (to prevent peripheral withdrawal effects)
* Patients treated with drugs metabolized by certain enzymes (CYP3A4 and P-gp)
* Patients with severe hepatic impairment
* Patients with end-stage renal disease
* Patients with heart failure
* Patients with severe dementia that impacts daily functioning
* Pregnant and lactating females
* Not postmenopausal females and of childbearing potential and not using an accepted method of birth control (i.e, surgical sterilization; intrauterine contraceptive device; oral contraceptive, diaphragm)
* Patients participated in another investigational drug or medical device study within 30 days of surgery or planning to be enrolled in another investigational drug or medical device study or any study in which active patient participation was required outside normal hospital data collection during the course of this study
* Patients deprived of liberty or placed under the authority of a tutor or curator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time of hospital discharge | Date at which treatment is initiated and date of hospital discharge (up to 12 days)
  Comparaison between treatment group and placebo group for post-operative length of stay between the date of hospital discharge and the date of surgery

SECONDARY OUTCOMES:
Rate of reinsertion of nasogastric tube | From post-surgery to hospital discharge (up to 12 days)
  Comparaison between treatment group and placebo group for rate of reinsertion of nasogastric tube
Time to reach gastrointestinal recovery | Date at which the patient has the first gaz from post-surgery (up to 12 days)
  Comparaison between treatment group and placebo group for time ot reach gastrointestinal recovery
Rate of 30-day postoperative complications | Postoperative complications from surgery, to 30-day postsurgery and to 90 postsurgery with Clavien-Dindo classification (up to 3 motnhs)
  Comparaison between treatment group and placebo group for rate of 30-day postoperative complications with Clavien-Dindo classification grade I-V
Rate of major postoperative complications of 90-day postoperative period | Major postoperative complications from surgery to 90 postsurgery with Clavien-Dindo classification (up to 3 motnhs)
  Comparaison between treatment group and placebo group for rate of major postoperative complications with Clavien-Dindo classification grade III-IV-V

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Pignot, MD, PhD, Principal Investigator — Isntitut Paoli-Calmettes